CLINICAL TRIAL: NCT01012219
Title: A Study to Evaluate the Effects of Laropiprant on the Antiplatelet Effects of Clopidogrel and Aspirin in Combination and to Evaluate Single Dose Pharmacokinetics of MK0524A in Subjects With Primary Hypercholesterolemia or Mixed Dyslipidemia
Brief Title: A Study to Evaluate the Effects of Laropiprant on the Antiplatelet Effects of Clopidogrel and Aspirin in Combination (MK-0524A-114)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-114; 2009_689
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Primary Hypercholesterolemia; Mixed Hyperlipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Niacin; MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Period 1 (Experimental): In Periods 1 and 2 each participant will receive one of the following treatments in a randomized crossover fashion: Treatment A (aspirin 81 mg, clopidogrel 75 mg and laropiprant 40 mg once daily for 7 days) or Treatment B (aspirin 81 mg, clopidogrel 75 mg and placebo to laropiprant 40 mg once daily for 7 days).
  Interventions: Drug: Comparator: aspirin; Drug: Comparator: clopidogrel; Drug: Comparator: laropiprant; Drug: Comparator: placebo
- Period 2 (Experimental): In Periods 1 and 2 each participant will receive one of the following treatments in a randomized crossover fashion: Treatment A (aspirin 81 mg, clopidogrel 75 mg and laropiprant 40 mg once daily for 7 days) or Treatment B (aspirin 81 mg, clopidogrel 75 mg and placebo to laropiprant 40 mg once daily for 7 days).
  Interventions: Drug: Comparator: aspirin; Drug: Comparator: clopidogrel; Drug: Comparator: laropiprant; Drug: Comparator: placebo
- Period 3 (Experimental)
  Interventions: Drug: niacin (+) laropiprant

INTERVENTIONS:
Drug: niacin (+) laropiprant — open-label, single dose Tredaptive (1000mg ER niacin/ 20mg laropiprant) 2 oral tablets
  Other Names: Tredaptive
  Arms: Period 3
Drug: Comparator: aspirin — 81 mg oral tablet once daily for 7 days
  Arms: Period 1; Period 2
Drug: Comparator: clopidogrel — 75 mg oral tablet once daily for 7 days
  Arms: Period 1; Period 2
Drug: Comparator: laropiprant — 40 mg oral tablet once daily for 7 days
  Arms: Period 1; Period 2
Drug: Comparator: placebo — placebo oral tablet once daily for 7 days
  Arms: Period 1; Period 2

SUMMARY:
This is a 3-period study. Periods 1 and 2 will evaluate the effects of multiple doses of laropiprant on the antiplatelet effects of clopidogrel and aspirin administered in combination in participants with primary hypercholesterolemia or mixed dyslipidemia. Period 3 will be open-label and will evaluate single dose pharmacokinetics of nicotinic acid and laropiprant components of Tredaptive.

ELIGIBILITY:
Inclusion Criteria:

* Participant has primary hypercholesterolemia or mixed dyslipidemia (high cholesterol)
* Participant is a non-smoker

Exclusion Criteria:

* Participant has a history of chronic seizures
* Participant has a history of cancer
* Participant has a history of stomach or intestinal ulcers or any history of GI bleeding
* Participant has had major surgery, donated blood or participated in another investigational study in the past 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] De Kam PJ, Luo WL, Wenning L, Ratcliffe L, Sisk CM, Royalty J, Radziszewski W, Wagner JA, Lai E. The effects of laropiprant on the antiplatelet activity of co-administered clopidogrel and aspirin. Platelets. 2014;25(7):480-7. doi: 10.3109/09537104.2013.836747. Epub 2013 Nov 8. PMID 24206527

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Periods 1 and 2 evaluated the effects of multiple doses of laropiprant on the antiplatelet effects of clopidogrel and aspirin administered in combination in participants with primary hypercholesterolemia or mixed dyslipidemia. Period 3 was open-label and evaluated single dose pharmacokinetics of nicotinic acid and laropiprant components of Tredaptive.
Period: Period 1
Arm/Group | All Participants
Started | 36 (Number randomized)
Completed | 35
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Period 2
Arm/Group | All Participants
Started | 35 (Number who completed Period 1)
Completed | 34
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Period 3
Arm/Group | All Participants
Started | 20 (of the 36 who started Period 1)
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: years] | 55.0 [24 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Cutaneous Bleeding Time (BT)
Description: Cutaneous bleeding Time (BT) on Day 8 after daily administration of laropiprant with aspirin and clopidogrel for 7 days versus BT on Day 8 after daily administration of placebo with aspirin and clopidogrel for 7 days.
  The model used included treatment, period and sequence as fixed effect variables and subjects as the random effect variable.
  Period 3 was not analyzed as bleeding time was not an objective for this part of the study.
Time Frame: Day 8
Population: Due to technical reasons, bleeding time was zero for some participants; they were considered to be missing data. Therefore, these observations were excluded from the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Seconds
Groups:
- Clopidogrel + Aspirin +Laropiprant; Clopidogrel + Aspirin: Participants from Periods 1 and 2
Arm/Group | Clopidogrel + Aspirin +Laropiprant | Clopidogrel + Aspirin
Number analyzed (Participants) | 34 | 33
Seconds | 478 [381 to 599] | 389 [309 to 490]
Statistical Analysis 1: Comparison: Clopidogrel + Aspirin +Laropiprant vs Clopidogrel + Aspirin; Test type: Superiority or Other; Geometric least-squares mean ratio = 1.23, 90% CI 2-sided [0.96 to 1.56]

ADVERSE EVENTS:
Groups:
- Laropiprant + Clopidrogel + Aspirin; Clopidogrel + Aspirin: Participants from Periods 1 and 2
- Laropiprant + Niacin: Participants from Period 3
Arm/Group | Laropiprant + Clopidrogel + Aspirin | Clopidogrel + Aspirin | Laropiprant + Niacin
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/20
Other Adverse Events (participants affected / at risk) | 24/36 | 23/36 | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Laropiprant + Clopidrogel + Aspirin (N=36) | Clopidogrel + Aspirin (N=36) | Laropiprant + Niacin (N=20)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 2 | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 6 | 3 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 2
Headache (Nervous system disorders) | 5 | 4 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 7 | 4 | 0
Flushing (Vascular disorders) | 2 | 0 | 0
Vasodilation (Vascular disorders) | 0 | 0 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.